CLINICAL TRIAL: NCT05016037
Title: Predictors of Speech Ability in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Stephen Camarata, Professor, Hearing and Speech Sciences, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Vanderbilt_UniversityMC; R21DC019280-01A1 (NIH)
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Speech Intelligibility Intervention in Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lexically Based Speech Intelligibility Recast (Other): Speech recasts are likely to improve speech intelligibility in Down Syndrome. The goal of this study is to induce change in speech intelligibility in order to study speech accuracy and prosody as predictors of change in speech intelligibility.
  Interventions: Behavioral: Lexically based speech recast

INTERVENTIONS:
Behavioral: Lexically based speech recast — A child's spontaneous or elicited word production containing phonological errors is immediately followed with a clinician verbal model that corrects the error(s) at the word level rather than the isolated phoneme level. As an example, a speech recast of child's production of the word "bake" as [be] would be the whole lexeme bake [bek] rather than production drill on [k] in isolation.
  Other Names: Phonological Recast

SUMMARY:
Speech is a critical aspect of the human experience and usually develops in a "seemingly automatic process that continues from birth through adolescence and underlies many related abilities" (e.g., language and reading, see National Academy of Medicine Report on Speech and Language Disorders, 2016). Many individuals with Down Syndrome (Trisomy 21, DS) struggle to communicate and participate more fully in human communication and educational learning experiences because their speech is difficult to understand. The purpose of the proposed project was to measure speech-articulation accuracy and speech intelligibility, and their proposed primary predictors at study entry in 16 children with DS age 4;0 to 17;11). A validated treatment, speech recast intervention (see Yoder, Camarata & Woynaroski, 2016) was used to drive growth in speech intelligibility as a means of evaluating changes in potential sequelae of change. This study included measures of speech-articulation accuracy, and speech-prosody skills as predictors of speech intelligibility growth in DS.

DETAILED DESCRIPTION:
In most children, speech development progresses in a "seemingly automatic manner that continues from birth through adolescence"1 and supports related communication and reading abilities. But many individuals with Down Syndrome (DS, about 1 in 700 births in the US) struggle to acquire speech and participate more fully in human communication and gain access to learning experiences, in part, because their speech is often difficult to understand. This persistent speech disorder arises because people with DS must acquire and produce speech using structurally-different articulators and poor speech oral-motor abilities. Moreover, there is considerable variability in the speech intelligibility of people with DS and it is unclear why some people with DS communicate relatively proficiently whereas others are unable to clearly communicate.

The Investigator's recent research provides a unique combination of findings that, when integrated into a prospective project, can potentially provide new insights into how people with DS improve speech intelligibility. This assertion is grounded in the long-standing and replicated finding that speech intelligibility in DS is not strongly correlated with nor solely attributable to measures of phoneme production, so that improvements in intelligibility must rely not only improvements in speech accuracy (phoneme production) but also upon changes in "nonphonemic" factors such as cognitive-linguistic parameters and suprasegmental features such as prosody and speech rate that are currently poorly understood. For example, in a recent paper (Wilson, Abedduto, Camarata & Shriberg, 2019), the Investigators describe cognitive/linguistic and speech-motor factors that relate to speech intelligibility in DS and provide preliminary data on nonphonemic parameters that are significantly correlated to intelligibility. In the cognitive linguistic domain, the Investigators found that measures of cognitive ability and receptive language abilities were directly related to speech intelligibility in people with DS. The Investigators also found that measures of speech-motor ability related to speech intelligibility. Importantly, in another series of studies, the Investigators demonstrated that individualized lexically based phonological recast intervention resulted in improvements in speech intelligibility in school age children with DS and that these gains were NOT uniquely attributable to changes in speech accuracy (phoneme production). Thus, the Investigators propose to induce growth in speech intelligibility in order to study change in speech and as an important step towards a) developing more effective speech interventions, and b) gaining a better understanding of parameters that drive improved speech intelligibility in DS (e.g.,phoneme production). This latter point is especially important because the Investigator's previous research and the extant literature indicate that traditional measures of speech accuracy (e.g., phoneme articulation) do not completely capture or predict improvements in speech intelligibility in DS. The proposed research would thus test assumptions underlying current models of speech disorder (and intervention) in DS. The Investigator's previous research has indicated that the Investigators can drive change in speech intelligibility without directly targeting speech accuracy, providing an opportunity to study intelligibility while controlling for speech accuracy as an untreated factor. Thus, an important first step in identifying factors that influence variation in speech intelligibility in addition to speech accuracy is to identify predictors of these speech abilities following intervention induced gains. Therefore, in keeping with the goals of an exploratory/developmental research project proposal (R21), the Investigators propose a pre-post design that measures speech intelligibility, and it's posited sequelae within the context of a controlled pre-post speech recast intervention study. Participants were 16 school-age children (4 to 17 years) with DS with varied cognitive ability levels (minimum of 60 with no ceiling). The following specific aims were pursued:

Aim 1: Test whether there were changes in baseline to post intervention measures of speech.

Aim 2: Examine the associations among measures of speech accuracy and prosody and overall speech intelligibility.

Impact: The results of this study within the context of a pre-post intervention design will provide important preliminary information on factors that contribute to intelligible speech in DS; thereby informing models of speech intelligibility and speech accuracy and future larger scale clinical trials. The proposed project will provide preliminary data to guide future longitudinal studies of value-added predictors of speech outcomes, and ultimately, improve assessment and intervention for speech deficits in individuals with DS.

ELIGIBILITY:
Inclusion Criteria:

* previous medical identification of Down Syndrome
* chronological age 4-17 years
* regular use of 3-word utterances (ascertained via parent report during screening and confirmed during assessments)
* pass a hearing screening at the time of enrollment in the project. All will pass a hearing screening (25 dB @1000, 2000, 4000 Hz).

Exclusion Criteria:

A history of or parent report of

* seizures,
* diagnosed ADHD,
* apraxia secondary to a diagnosed neurological disorder
* Autism Spectrum Disorder (Autism Diagnostic Observation Scale-2nd Edition score above the ASD cut-off) or
* severe disruptive behavior that would prevent participation in testing or treatment.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Camarata, PhD, Principal Investigator — VUMC Dept of Hearing & Speech Sciences
Locations (1):
- VUMC Bill Wilkerson Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoder PJ, Camarata S, Woynaroski T. Treating Speech Comprehensibility in Students With Down Syndrome. J Speech Lang Hear Res. 2016 Jun 1;59(3):446-59. doi: 10.1044/2015_JSLHR-S-15-0148. PMID 27300156
- [Background] Yoder PJ, Woynaroski T, Camarata S. Measuring Speech Comprehensibility in Students with Down Syndrome. J Speech Lang Hear Res. 2016 Jun 1;59(3):460-7. doi: 10.1044/2015_JSLHR-S-15-0149. PMID 27299989
- [Background] Wilson EM, Abbeduto L, Camarata SM, Shriberg LD. Speech and motor speech disorders and intelligibility in adolescents with Down syndrome. Clin Linguist Phon. 2019;33(8):790-814. doi: 10.1080/02699206.2019.1595736. PMID 31221010

RESULTS

PARTICIPANT FLOW:
Groups:
- Lexically Based Speech Intelligibility Recast: Speech recasts are likely to improve speech intelligibility in Down Syndrome. The goal of this study is to induce change in speech intelligibility in order to study phonological, acoustic and suprasegmental sequelae of improvements in speech.
  Lexically based speech recast: a child's spontaneous or elicited production containing phonological errors is immediately followed with a clinician model that corrects the error(s) at the word level rather than the isolated phoneme level. As an example, a speech recast of child's production of the word bake as [be] would be the whole lexeme bake [bek] rather than production drill on [k] in isolation.
Period: Overall Study
Arm/Group | Lexically Based Speech Intelligibility Recast
Started | 18
Completed | 16
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: 18 participants signed informed consent. One person did not complete the baseline assessment and withdrew from the study.
Groups:
- Baseline Measures: Baseline Measures and Demographic Information
Arm/Group | Baseline Measures
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17
Leiter International Performance Scale, Third Edition [Mean (Standard Deviation); unit: Nonverbal IQ] — The Leiter International Performance Scale, Third Edition measures nonverbal IQ across four subscales, including Sequential Order (SO), Form Completion (FC), Classification and Analogies (CA), and Figure Ground (FG). Nonverbal IQ scores range is 30-170, which encompass 'severe delay' to 'extremely high/gifted', higher numbers indicates higher intelligence.
  Nonverbal IQ | 71.69 (13.26)
Receptive One Word Picture Vocabulary Test (ROWPVT-4) [Mean (Standard Deviation); unit: Standard Score] — The Receptive One Word Picture Vocabulary Test (ROWPVT-4) is a measure of word understanding. The test includes 190 items (correct or incorrect). Knowledge of receptive vocabulary is measured by asking the respondent to point to one of four pictures that corresponds to a word (object, person, or action) spoken by the assessor. Scores range from 0-190, with higher scores denoting better performance relative to same age peers.
  Standard Score | 74.75 (13.42)
Expressive One Word Picture Vocabulary Test (EOWPVT-4) [Mean (Standard Deviation); unit: standard score] — The Expressive One Word Picture Vocabulary Test (EOWPVT-4) is a measure of expressive vocabulary. The test includes 190 items (correct or incorrect) used to assess children's ability to verbally label illustrations of objects, actions, or concepts. Knowledge of expressive vocabulary is measured by the assessor pointing to a picture and the child naming it. Scores range from 0 to 190. Higher scores denote better performance relative to same age peers.
  standard score | 73.7 (10.5)
Arizona Articulation and Phonology Scale-4th Edition [Mean (Standard Deviation); unit: Standard Score] — The Arizona Articulation and Phonology Scale-4th Edition (Arizona-4) evaluates articulatory and phonological skills. 43 pictures are used to measure correctly produced speech sounds as expressed in the production of 43 single words (Word Articulation Test). The same 43 single words in the Word Articulation test are embedded into sentences to measure articulatory ability in the Sentence Articulation Test. Combined scores from the 2 tests range from 0-86. Higher scores denote stronger skills.
  Standard Score | 57.5 (2.1)
Woodcock Camarata Articulation Battery (WCAB) [Mean (Standard Deviation); unit: standard score] — Woodcock Camarata Articulation Battery (WCAB) is a rating of word intelligibility. The test includes 67 items each scored as correct or incorrect. Scores range from 0-67. Higher scores denote better word intelligibility.
  standard score | 32.56 (15.43)
Test for Auditory Comprehension of Language - 4th Edition (TACL-4) [Mean (Standard Deviation); unit: standard score] — The TACL-4 assesses a child's receptive spoken language abilities among 3 subtests: Vocabulary, Grammatical Morphemes, and Elaborated Phrases and Sentences. 142 stimulus items each have a corresponding picture plate with 3 colored drawings. Participants point to the picture that best represents the meaning of the stimulus. The raw score is the total number of correct responses, applying basal (3 correct answers) & ceiling (3 incorrect answers) rules to each subtest to determine the number of items administered and scored. Scores range from 0-142. Higher scores denote greater language ability.
  standard score
    Vocabulary Subtest | 52.06 (24.74)
    Grammatical Morphemes | 47.12 (16.6)
    Elaborated Phrases and Sentences | 46.56 (15.66)
Percent Consonants Correct [Median (Standard Deviation); unit: Percent Consonants Correct] — Percent Consonants Correct is a measure of the percentage of consonants correctly produced on the Arizona Articulation and Phonology Scale-4th Edition.
  Percent Consonants Correct | 61.81 (20.45)
Percent Vowels Correct [Mean (Standard Deviation); unit: Percent Vowels Correct] — Percent Vowels Correct is a measure of the percentage of vowels correctly produced on the Arizona Articulation and Phonology Scale-4th Edition.
  Percent Vowels Correct | 88.82 (9.37)
Mean Length of Utterance [Mean (Standard Deviation); unit: morphemes per phrase] — Mean Length of Utterance is the average number of morphemes in each phrase that are correctly produced during a spontaneous language sample
  morphemes per phrase | 2.24 (1.17)
Speech Intelligibility [Mean (Standard Deviation); unit: score on a scale] — Speech intelligibility is a 5 point Likert scale based on the language sample obtained (e.g., based on the number of words spoken in the sample). The scale range is 1 to 5, 1 being very low intelligibility and 5 being high intelligibility.
  score on a scale | 3.53 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: Speech Intelligibility
Description: Speech intelligibility is a 5 point Likert scale based on the language sample obtained (e.g., based on the number of words spoken in the sample). The scale range is 1 to 5, 1 being very low intelligibility and 5 being high intelligibility.
Time Frame: six months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lexically Based Speech Intelligibility Recast: School-age children (4-17 years) with Downs Syndrome with varied cognitive ability levels (minimum of 60 with no ceiling)
Arm/Group | Lexically Based Speech Intelligibility Recast
Number analyzed (Participants) | 16
score on a scale | 3.59 (0.97)

2. Primary Outcome: Speech Accuracy
Description: Percentage of correct phonemes on standardized speech tests and in a semi structured speech sample. This is the number of correct phonemes divided by the number of total phonemes in the sample (or test) divided by 100.
Time Frame: six months
Population: One participant did not complete the final speech accuracy measure. The patient declined (refused) to complete the test. The assent rules require that the study team stop testing if a child indicates they do not want to do a test.
Measure: Mean (Standard Deviation); unit: percentage of correct phonemes
Arm/Group | Lexically Based Speech Intelligibility Recast
Number analyzed (Participants) | 15
percentage of correct phonemes
  Percent Consonants Correct | 61.55 (17.97)
  Percent Vowels Correct | 89.57 (9.05)

ADVERSE EVENTS:
Time Frame: Participants were enrolled in the study for ~ 6 months long (from Baseline assessments to Post assessments)
Arm/Group | Lexically Based Speech Intelligibility Recast
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
Limitations include that there is no control group, therefore results are not evidence of the efficacy/efficiency of lexical recast intervention on speech production in children with Down syndrome (DS). A caveat is the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT05016037/Prot_001.pdf
  • Statistical Analysis Plan (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT05016037/SAP_002.pdf
  • Informed Consent Form (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT05016037/ICF_003.pdf